CLINICAL TRIAL: NCT03809442
Title: Analgesic Efficacy of Ropivacaine Alone or in Combination With Adjuvants on Post-operative Analgesia Following Video-Assisted Thoracoscopic Surgery (VATS) - A Randomized Controlled Trial.
Brief Title: Analgesic Efficacy of Ropivacaine Alone or in Combination With Adjuvants on Post-operative Analgesia Following Video-Assisted Thoracoscopic Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Saad Yousuf, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0743
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Ropivacaine; Ketamine; Tramadol; Midazolam; Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Ropivacaine with Ketamine (Experimental): Ropivacaine is a propyl analog of bupivacaine with longer duration of action with much safer cardiotoxicity profile than bupivacaine. Ropivacaine has the same analgesic effects as bupivacaine and levobupivacaine, but it is associated with a low incidence of motor block. Thus, ropivacaine appears to be an important component for local anesthesia and postoperative analgesia.
  Ketamine is an N-methyl-D-aspartate (NMDA) receptor antagonist that possesses both central and peripheral analgesic effects. Preincisional infiltration of ketamine prolongs the time to first analgesic requirement and also decreases the total amount of analgesics used postoperatively.
  Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 1mg/kg ketamine (8 mL per incision) (ketamine group).
  Interventions: Drug: Ropivacaine + Ketamine
- Ropivacaine with Tramadol (Experimental): Tramadol hydrochloride is a synthetic analog of codeine that acts on both opioid (weak mu receptor agonist) and nonopioid receptors (inhibits reuptake of nor-adrenaline and serotonin as well as release stored serotonin from nerve endings) which play a crucial role in pain inhibition pathway.
  It also blocks nerve conduction which imparts its local anesthetics like action on peripheral nerves.
  In one study it was found that the addition of tramadol or midazolam to caudal epidural ropivacaine prolongs the duration of analgesia without causing significant side effects.
  Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 2mg/kg tramadol (8 mL per incision) (Tramadol group).
  Interventions: Drug: Ropivacaine + Tramadol
- Ropivacaine with Midazolam (Experimental): The analgesic effect of extradurally administered midazolam is through γ-amino butyric acid (GABA)/benzodiazepine system of spinal cord.
  Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 50 μg/kg midazolam (8 mL per incision) (Midazolam group).
  Interventions: Drug: Ropivacaine + Midazolam
- Ropivacaine with Dexamethasone (Experimental): The glucocorticoid dexamethasone appears to be effective in a small number of preclinical and clinical studies and found that dexamethasone prolongs analgesia from interscalene blocks using ropivacaine or bupivacaine, with the effect being stronger with ropivacaine.
  Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine+ 8mg dexamethasone (8 mL per incision) (Dexamethasone group).
  Interventions: Drug: Ropivacaine + Dexamethasone
- Ropivacaine with Dexmedetomidine (Experimental): Dexmedetomidine is a new highly selective alpha2 (a2) agonist with known sedative, antihypertensive, anxiolytic, and analgesic properties.
  In one study, it was found that wound infiltration with combined ropivacaine and dexmedetomidine found to be significantly superior for postoperative analgesia compared with either combined ropivacaine and tramadol or ropivacaine alone for lumbar discectomies.
  Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% Ropivacaine + 0.5μg/kgdexmedetomidine (8mL per incision) (Dexmedetomidine group).
  Interventions: Drug: Ropivacaine + Dexmedetomidine
- Ropivacaine (Placebo Comparator): Ropivacaine is a propyl analog of bupivacaine with longer duration of action with much safer cardiotoxicity profile than bupivacaine. Ropivacaine has the same analgesic effects as bupivacaine and levobupivacaine, but it is associated with a low incidence of motor block. Thus, ropivacaine appears to be an important component for local anesthesia and postoperative analgesia.
  Patients will receive subcutaneous wound infiltration with 24ml of 0.25% Ropivacaine in three divided doses (i.e. 8 mL per incision) (control group). Total dose of Ropivacaine will be 60 mg.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine + Ketamine — Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 1mg/kg ketamine (8 mL per incision) (ketamine group).
  Arms: Ropivacaine with Ketamine
Drug: Ropivacaine + Tramadol — Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 2mg/kg tramadol (8 mL per incision) (Tramadol group).
  Arms: Ropivacaine with Tramadol
Drug: Ropivacaine + Midazolam — Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 50 μg/kg midazolam (8 mL per incision) (Midazolam group).
  Arms: Ropivacaine with Midazolam
Drug: Ropivacaine + Dexmedetomidine — Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% Ropivacaine + 0.5μg/kg dexmedetomidine (8mL per incision) (Dexmedetomidine group).
  Arms: Ropivacaine with Dexmedetomidine
Drug: Ropivacaine + Dexamethasone — Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine+ 8mg dexamethasone (8 mL per incision) (Dexamethasone group).
  Arms: Ropivacaine with Dexamethasone
Drug: Ropivacaine — Patients will receive subcutaneous wound infiltration with 24ml of 0.25% Ropivacaine in three divided doses (i.e. 8 mL per incision) (control group). Total dose of Ropivacaine will be 60 mg.
  Arms: Ropivacaine

SUMMARY:
The aim of the study is to investigate the analgesic effects of the subcutaneous wound infiltration with tramadol, ketamine, dexamethasone, dexmedetomidine and midazolam as adjuvant to ropivacaine, compared to ropivacaine alone in patients undergoing Video-Assisted thoracoscopic Surgery (VATS) procedures.

DETAILED DESCRIPTION:
After obtaining approval from Ethical Review Committee (ERC) of Aga Khan University Hospital Karachi (AKUH), and inform about the study to primary surgeon, informed written consent will be obtained from the patients fulfilling the inclusion criteria.

Patients will be recruit in the study during the preoperative anesthesia evaluation either at the preoperative clinic or from the ward after admission. Their Medical Record (MR) number will be send to the Clinical Trials Unit (CTU), along with their expect date, day and timing of surgery. The CTU will randomly allocate the patients to one of the six groups, based on computer generated allocation. After the patient will reach the preoperative area in the operating room (OR), an email request will be generated to the CTU who will release the prepared study drug syringe and will send it to the Principal Investigator (PI). The syringe contain either Ropivacaine alone or in combinations with other adjuvants. The drugs for all six groups looks alike, so that the patient, principal investigator, and surgeon administering the drugs or making observations will all blinded.

Group A: Patients will receive subcutaneous wound infiltration with 24ml of 0.25% Ropivacaine in three divided doses (i.e. 8 mL per incision) (control group). Total dose of Ropivacaine will be 60 mg.

Group B: Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 1mg/kg ketamine (8 mL per incision) (ketamine group).

Group C: Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 2mg/kg tramadol (8 mL per incision) (Tramadol group).

Group D: Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine + 50 μg/kg midazolam (8 mL per incision) (Midazolam group).

Group E: Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% ropivacaine+ 8mg dexamethasone (8 mL per incision) (Dexamethasone group).

Group F: Patients will receive subcutaneous wound infiltration with total volume of 24 mL of 0.25% Ropivacaine + 0.5μg/kg dexmedetomidine (8mL per incision) (Dexmedetomidine group).

All patient will be given general anesthesia as per standard of care. Subjects will be blinded to the identity of the study drug they receive for postoperative analgesia. The study drugs will be prepared by an anaesthesiologist unrelated to the study and will be infiltrated by the surgeon intraoperatively before skin closure.

Pre-operatively, patients will be taught how to evaluate pain intensity using the visual analogue scale (VAS) scored from 0 to 10 (where 0 = no pain and 10 = worst pain).On arrival to the operative room, routine monitoring including ECG, non-invasive blood pressure, pulse oximetry and capnography was applied. All patient will be pre-medicated with tablet midazolam 7.5mg PO before surgery.

In all patients, general anaesthesia will be induce with intravenous morphine (0.1mg/kg) and 2 mg/kg propofol; endotracheal intubation will be facilitated with 0.5 mg/kg atracurium. Anaesthesia will be maintain with inhalational anaesthetic (MAC 1.2 -1.4%) isoflurane in 50% oxygen/air mixture and 0.03 mg/kg atracurium bolus given every 30 min. Intraoperatively, intravenous paracetamol (15mg/kg) will be given to all patients. In Video assisted thoracotomy surgery (VATS), three incision lines are used for port insertion. Surgeries which involves less than 3 ports will be excluded. Just before skin closure, surgeon will infiltrate the prepared study drug (groups will be randomly allocated preoperatively), 8 ml per incision site. Prophylactic antiemetic (Ondansetron 4 mg) will be given intraoperatively.

Postoperatively, all patients will admit to postanaesthesia care unit (PACU); the patients' heart rate, non-invasive blood pressure, respiratory rate and oxygen saturation will be monitor and record. The presence and severity of pain at rest(VAS-R) and on coughing (VAS-M) will be assess by using VAS score, and sedation will be assess by using sedation score as (awake and alert = 0, quietly awake = 1, asleep but easily aroused = 2, deeply asleep = 3) at the following time points: at 0, 2, 6, 12 and 24 h postoperatively. The time to first request for rescue analgesia will be recorded Patients will be given tramadol 50mg intravenously (as per need) upon request for initial rescue analgesia (if VAS score >4), which then will be given on regular doses (tramadol 50 mg IV every 8 hourly along with paracetamol 1 gm IV every 6 hourly).

Adverse effects:

Adverse Events are defined as 'Any untoward medical occurrence in a trial patient to whom a research treatment or procedure has been administered, including occurrences which are not necessarily caused by or related to that treatment or procedure.

Post-operative assessment of other effects patients will be observed any of the following till 2 hours to discharge of the patient from PACU.

* Hallucination is a sensory perception experienced in the absence of an external stimulus as distinct from an illusion which is a misperception of an external stimulus.
* Nystagmus is rapid involuntary rhythmic eye movement, with the eyes moving quickly in one direction (quick phase), and then slowly in the other (slow phase).
* Nausea is the sensation of unease and discomfort in the stomach with an urge to vomit.
* Sedation is define as, reduction of anxiety, stress, irritability, or excitement
* Respiratory depression (Respiratory rate less than 8/min)
* Hypo and hypertension (Systolic blood pressure <90 mm Hg or > 140 mm Hg)

Management of side effects:

* If hallucination or nystagmus happens, then it will be manage by giving intravenous haloperidol 5mg and observe the patient.
* If patient complains of nausea, it will be manage by giving intravenous injection metoclopramide 10mg
* If respiratory depression happens, then it will be manage by titrating the amount of injection naloxone 0.1mg intravenously and monitor the patient.
* If hypotension happen, then it will be manage by giving intravenous fluid and see the response, if hypotension persists then investigator will give injection ephedrine or phenylephrine in titrating dose.
* If hypertension occurs, it will be manage by giving intravenous hydralazine or metoprolol in titrating dose.

Serious Adverse Events:

* Serious Adverse Events are defined as an untoward event that: Results in death; Is life-threatening*; Requires hospitalization** or prolongation of existing hospitalization; Results in persistent or significant disability or incapacity; Or, is otherwise considered medically significant by the Investigator (18)
* *The term "life-threatening" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe. ** Patients must be formally admitted - waiting in out-patients or A&E does not constitute an SAE (even though this can sometimes be overnight). Similarly, planned hospitalizations that clearly are not related to the condition under investigation or hospitalizations/prolongation of hospitalization due to social reasons should not be considered as serious adverse event (18).

There is no direct financial or other benefit for the participant of the study. However, these medicines will be provided free. In case of any event related to the study drug, it will be managed & cost will be borne by the institution.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I to III.
2. Age >18 years.
3. Either sex.
4. Elective Video assisted thoracotomy surgery (VATS) under general anaesthesia

Exclusion Criteria:

1. ASA IV & V.
2. Coagulation disorders.
3. Infection at the vicinity of the surgical wound.
4. Raised intracranial pressure.
5. History of hypersensitivity or known allergy to any study drug.
6. History of opioid addiction.
7. History of seizure disorder.
8. Those who are not willing to participate in the study.
9. Allergy to local anesthetics.
10. Duration of surgery greater than 2 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Time to the first postoperative analgesia requirement | Follow till 24 hours postoperatively
  Time to the first analgesic requirement will be calculated as the time from the performance of local wound infiltration to the first analgesic dose administered. This time will be noted in minutes.
Visual analogue scale (VAS) | Follow till 24 hours postoperatively
  Assessement for Postoperative Pain.
  The requirement of postoperative analgesia of the patient will be evaluated by using Visual analogue scale (VAS). It scored from 0 to 10 (where 0 [minimum score] = no pain and 10 [maximum score] = worst pain). Aggregate score will be added.
  Score less than 4 will be consider adequate analgesia while score greater than 4 will be consider inadequate analgesia. This score is just a numerical number with no other value attached to it.

SECONDARY OUTCOMES:
Sedation using Pasero Opioid-Induced Sedation Scale (POSS) | Follow till 24 hours postoperatively
  Sedation will be assessed by using Pasero Opioid-Induced Sedation Scale (POSS).
  This scale measures sedation on numerical score of 0 to 4. Minimum score is 0 while maximum score is 4.
  It comprises of; 0: awake; 1: mild sedation; 2: sleeping, but able to wake; 3: Frequently drowsy, arousable, drifts off to sleep during conversation, unable to wake and 4: Somnolent, minimal or no response to verbal or physical stimulation.
  A POSS score of 0, 1, or 2 indicates an acceptable level of sedation, whereas a score of 3 or 4 indicates over-sedation and the need for a reversal agent.
  This score is just a numerical number with no other value attached to it.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sommer M, de Rijke JM, van Kleef M, Kessels AG, Peters ML, Geurts JW, Gramke HF, Marcus MA. The prevalence of postoperative pain in a sample of 1490 surgical inpatients. Eur J Anaesthesiol. 2008 Apr;25(4):267-74. doi: 10.1017/S0265021507003031. Epub 2007 Dec 6. PMID 18053314
- [Background] Bernucci F, Carli F. Functional outcome after major orthopedic surgery: the role of regional anesthesia redefined. Curr Opin Anaesthesiol. 2012 Oct;25(5):621-8. doi: 10.1097/ACO.0b013e328357a3d5. PMID 22914354
- [Background] Bafna U, Sharma G, Sapru S, et al. Comparison of clonidine anddexmedetomidine as an adjuvant to 0.5% ropivacaine in supraclavicularbrachial plexus block: a prospective, randomized,doubleblindand controlled study. J Recent Adv Pain. 2015;1:73-77.
- [Background] Ng A, Swami A, Smith G, Davidson AC, Emembolu J. The analgesic effects of intraperitoneal and incisional bupivacaine with epinephrine after total abdominal hysterectomy. Anesth Analg. 2002 Jul;95(1):158-62, table of contents. doi: 10.1097/00000539-200207000-00028. PMID 12088961
- [Background] Li M, Wan L, Mei W, Tian Y. Update on the clinical utility and practical use of ropivacaine in Chinese patients. Drug Des Devel Ther. 2014 Sep 9;8:1269-76. doi: 10.2147/DDDT.S57258. eCollection 2014. PMID 25246768
- [Background] Pedersen JL, Galle TS, Kehlet H. Peripheral analgesic effects of ketamine in acute inflammatory pain. Anesthesiology. 1998 Jul;89(1):58-66. doi: 10.1097/00000542-199807000-00011. PMID 9667294
- [Background] Tan PH, Cheng JT, Kuo CH, Tseng FJ, Chung HC, Wu JI, Hsiao HT, Yang LC. Preincisional subcutaneous infiltration of ketamine suppresses postoperative pain after circumcision surgery. Clin J Pain. 2007 Mar-Apr;23(3):214-8. doi: 10.1097/AJP.0b013e31802e3377. PMID 17314579
- [Background] Lewis KS, Han NH. Tramadol: a new centrally acting analgesic. Am J Health Syst Pharm. 1997 Mar 15;54(6):643-52. doi: 10.1093/ajhp/54.6.643. PMID 9075493
- [Background] Desmeules JA, Piguet V, Collart L, Dayer P. Contribution of monoaminergic modulation to the analgesic effect of tramadol. Br J Clin Pharmacol. 1996 Jan;41(1):7-12. doi: 10.1111/j.1365-2125.1996.tb00152.x. PMID 8824687
- [Background] Krishnadas A, Suvarna K, Hema VR, Taznim M. A comparison of ropivacaine, ropivacaine with tramadol and ropivacaine with midazolam for post-operative caudal epidural analgesia. Indian J Anaesth. 2016 Nov;60(11):827-832. doi: 10.4103/0019-5049.193672. PMID 27942056
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Reddy VS, Shaik NA, Donthu B, Reddy Sannala VK, Jangam V. Intravenous dexmedetomidine versus clonidine for prolongation of bupivacaine spinal anesthesia and analgesia: A randomized double-blind study. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):342-7. doi: 10.4103/0970-9185.117101. PMID 24106359
- [Background] Mitra S, Purohit S, Sharma M. Postoperative Analgesia After Wound Infiltration With Tramadol and Dexmedetomidine as an Adjuvant to Ropivacaine for Lumbar Discectomies: A Randomized-controlled Clinical Trial. J Neurosurg Anesthesiol. 2017 Oct;29(4):433-438. doi: 10.1097/ANA.0000000000000422. PMID 28266950